CLINICAL TRIAL: NCT01738412
Title: Validation of an Electroencephalograph Based Algorithm for Detection of Onset and Deterioration of Acute Ischemic Stroke by Comparison to NIHSS.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Neurokeeper Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: NK-002
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Stroke
Keywords: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study population: Stroke patients
  Interventions: Device: Neurokeeper stroke detector

INTERVENTIONS:
Device: Neurokeeper stroke detector — Monitoring stroke patients

SUMMARY:
The purpose of this study is the validation of an Electroencephalograph based algorithm for detection of onset and deterioration of Acute Ischemic Stroke by Comparison to NIHSS.

DETAILED DESCRIPTION:
Inclusion criteria study population

1. Age > 18 years old.
2. Acute stroke symptoms onset within 2 weeks of inclusion, and as proximate to event as possible and as long as there was no neurological deterioration (ΔNIHSS>4) from symptoms onset to inclusion.
3. Patients with TIA lasting at least 5 minutes or minor acute ischemic stroke (NIHSS < 4 at the time of enrolment)
4. More than 3 of the following:

Blood pressure >140/90 or unknown, Irregular heartbeat, Atrial Fibrillation, Smoker, Cholesterol >240 or unknown, Has Diabetes, Lack of physical exercise, Overweight, Has Stroke in the family

OR between 4 and 6 of the following:

Blood pressure 120-139/80-89, Unknown Irregular heartbeat, Atrial Fibrillation, Trying to quit smoking, Cholesterol 200-239, Borderline Diabetes, Some exercise, Slightly overweight, Not sure if Stroke occurred in family

Exclusion criteria study population

1. Intracranial hemorrhage on admission by CT.
2. Previous major hemispheric stroke.
3. Patients with pure sensory symptoms,
4. Significant movement disorder.
5. Local skull or skin affliction which prevents sensor application.
6. Any known condition which in the opinion of the investigator may interfere with the protocol implementation.

ELIGIBILITY:
Inclusion criteria study population

1. Age > 18 years old.
2. Acute stroke symptoms onset within 2 weeks of inclusion, and as proximate to event as possible and as long as there was no neurological deterioration (ΔNIHSS>4) from symptoms onset to inclusion.
3. Patients with TIA lasting at least 5 minutes or minor acute ischemic stroke (NIHSS < 4 at the time of enrolment)
4. More than 3 of the following:

Blood pressure >140/90 or unknown, Irregular heartbeat, Atrial Fibrillation, Smoker, Cholesterol >240 or unknown, Has Diabetes, Lack of physical exercise, Overweight, Has Stroke in the family

OR between 4 and 6 of the following:

Blood pressure 120-139/80-89, Unknown Irregular heartbeat, Atrial Fibrillation, Trying to quit smoking, Cholesterol 200-239, Borderline Diabetes, Some exercise, Slightly overweight, Not sure if Stroke occurred in family

Exclusion criteria study population

1. Intracranial hemorrhage on admission by CT.
2. Previous major hemispheric stroke.
3. Patients with pure sensory symptoms,
4. Significant movement disorder.
5. Local skull or skin affliction which prevents sensor application.
6. Any known condition which in the opinion of the investigator may interfere with the protocol implementation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)

PRIMARY OUTCOMES:
Detection of stroke
  EEG base algorithm system to detect and monitor changes in cerebral electrophysiological parameters as compared to clinical evaluation as assessed by NIHSS score.

SECONDARY OUTCOMES:
Correlation to severity of stroke
  Correlations between EEG + ERP changes and clinical status as assessed by NIHSS score.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel